CLINICAL TRIAL: NCT04715451
Title: A Novel Swaddling Method To Improve Developmental Care for Preterm Babies
Brief Title: Swaddling to Improve Neurodevelopment for Preterm Babies
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn due to staffing/funding concerns.
Sponsor: Johns Hopkins University (Other)
Collaborators: The Thomas Wilson Sanitarium for Children of Baltimore City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00261157
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Preterm Birth; Neurodevelopmental Disorders
Keywords: Preterm; Brain; Neurodevelopment; Swaddling
MeSH Terms: conditions — Premature Birth; Neurodevelopmental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Swaddle (No Intervention): The management of the non-intervention group is with a cotton swaddle that is standard of care. It represents a conventional standard management method using a swaddle made of cotton.
- Novel Swaddle (Experimental): The Novel Swaddle is made of fabric consisting of 85% nylon and 15% polyurethane. This fabric provides heat retention, is hygroscopic and stretches in both longitudinal and transverse directions, thus more accurately replicating the intrauterine environment. The novel material is sewed into a bag shape.
  Interventions: Other: Novel Swaddle

INTERVENTIONS:
Other: Novel Swaddle — A novel swaddling method.
  Arms: Novel Swaddle

SUMMARY:
The investigators will test a new medical grade swaddling system for optimal and more appropriate positioning for preterm infants. This is a trial focused on sleep state, state regulation and long-term neurodevelopment. The central hypothesis is that this novel swaddling method will promote sleep and an optimal sleep-wake cycle, while also improving the neurodevelopment of preterm infants. It is proposed that adequate positioning and secondary feedback of natural movement of arms and legs stimulates and fosters normal brain development.

DETAILED DESCRIPTION:
Throughout pregnancy, the fetus is encouraged to develop by maintaining proper flexed posture in the uterus and freely moving its arms and legs against the flexible boundaries of the womb. However, when born too early, preterm infants lose the natural boundaries of the womb that support this flexor positioning and movement support. In addition preterm infants undergo stress because of essential treatments in neonatal intensive care units and exposure to the extrauterine environment. To support the development of preterm infants, cotton wraps are often used to maintain appropriate body positioning. Swaddling helps maintain continuous and adequate body positioning which aids and provides a stable sleep environment and encourages muscle tone. However, traditional swaddling is challenging in preterm infants and preterm infants frequently become unswaddled. It is fraught with difficulties related to the neonatal care and monitoring preterm infants receive due to the prematurity. In addition, this stiff material does not provide the same sensory experience as the flexible boundaries of the womb. In response to this challenge, The Investigators developed a new medical grade swaddling system for optimal and more appropriate positioning and natural movement. Here, The Investigators outline a trial focused on sleep state, state regulation and long-term neurodevelopment. The central hypothesis is that this novel swaddling method will promote sleep and an optimal sleep-wake cycle, while also improving the neurodevelopment of preterm infants. It is proposed that adequate positioning and secondary feedback of natural movement of arms and legs stimulates and fosters normal brain development. The Investigators will clinically evaluate sleep at the level of amplitude-integrated electroencephalograph (aEEG) activity and perform the Prechtl's Assessment of General Movements (GMA) to assess spontaneous writhing and fidgety movements, which predicts the future neurodevelopment of preterm babies. The Investigators will also perform the Neonatal Intensive Care Unit (NICU) Network Neurobehavioural Scale (NNNS) as a standardized assessment of neurological integrity and organization. The goal is to provide early intervention to improve development in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Born very preterm (<32 weeks postmenstrual age (PMA))
* At least 12 hours and less than 2 months old
* Expected to survive > 3 days
* No congenital anomaly or genetic disorder with expected survival less than term equivalent
* No malformations requiring surgery within 1 month of life
* Central intravenous lines removed
* Approval of the primary neonatologist, ideally not a study team member, to approach family for consent
* Appropriate parent or guardian to provide informed consent

Exclusion Criteria:

* Life expectancy < 3 days
* Severe congenital anomaly or genetic disorder with life expectancy <40 weeks PMA
* Seizures
* Need for seizure medication
* Hypertension for age requiring medication
* Severe hematologic crisis such as disseminated intravascular coagulation
* Hydrops fetalis
* Clinical concern or diagnosis of toxoplasmosis, cytomegalovirus rubella or syphilis infection
* Clinical concern or diagnosis of severe acute respiratory distress syndrome coronavirus 2 (SARS CoV-2) or coronavirus disease (COVID-19)
* Central intravenous access and reliance on parenteral nutrition >50%
* Respiratory support greater than nasal canulae or nasal continuous positive airway pressure (CPAP) (i.e. ventilator dependent)
* Active infection, including need for antibiotics greater than 5 days (i.e. confirmed infection)
* Complex congenital heart disease
* Known chromosomal abnormalities
* Clinical or echocardiographic signs of symptomatic pulmonary hypertension
* Profound perinatal hypoxia-ischemia
* Receiving treatment for pain control
* Sustained tachypnea >80 breaths/minute
* Need for volume expansion or administration of inotropes
* No one available or willing to provide consent

Ages: 24 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-04-21 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
Change in Sleep-Wake Cycling Maturity as assessed by amplitude integrated EEG (aEEG) readings | 32 weeks postmenstrual age, 34 weeks postmenstrual age and 36 weeks postmenstrual age
  Using aEEG, the Investigators will assess the presence or absence of mature sleep-wake cycling as defined as regular rhythmic sinusoidal variations of amplitude with a cycle greater than or equal to 20 minutes. Tracings with a cycling pattern that does not fit into a mature sleep-wake cycle for the majority of the tracing will be classified as intermediate.
Change in length of time spent in sleep | 32 weeks postmenstrual age, 34 weeks postmenstrual age and 36 weeks postmenstrual age
  Using aEEG, the Investigators will assess the change in length of time (in minutes) spent in sleep.
Change in the number of awakenings in a 3 hour time period | 32 weeks postmenstrual age, 34 weeks postmenstrual age and 36 weeks postmenstrual age
  Using aEEG, the Investigators will assess the change in number of awakenings in a 3 hour time period.
Change in voltage as assessed by aEEG) readings | 32 weeks postmenstrual age, 34 weeks postmenstrual age and 36 weeks postmenstrual age
  Using aEEG, the Investigators will assess the change in voltage (measured in microvolts).
Change in ratio of active sleep and quiet sleep as assessed by amplitude integrated EEG (aEEG) readings | 32 weeks postmenstrual age, 34 weeks postmenstrual age and 36 weeks postmenstrual age
  Using aEEG The Investigators will assess the time spent in active sleep (irregular and low in amplitude) and quiet sleep (regular and high in amplitude).
Change in Sleep-Wake Cycling Continuity as assessed by amplitude integrated EEG (aEEG) readings | 32 weeks postmenstrual age, 34 weeks postmenstrual age and 36 weeks postmenstrual age
  Using aEEG The Investigators will examine the background activity on recordings to assess the presence or absence of isoelectric periods along with amplitude fluctuations. Tracings will be classified as continuous, discontinuous and borderline.

SECONDARY OUTCOMES:
Behavioral Maturity as assessed by the NNNS | 37 weeks postmenstrual age
  The NICU Network Neurobehavioural Scale (NNNS) is a standardized clinical assessment tool used to assess neurological integrity and organization in a single, structured clinical exam. Summary scores are created for neurobehavioral domains including: habituation, attention, handling, quality of movement, self-regulation, non optimal reflexes, asymmetrical reflexes, stress/abstinence, arousal, hypertonicity, excitability, and lethargy. 13 summary scores will be generated.
Change in General Movements as assessed by the GMA | 32 weeks postmenstrual age and 37 weeks postmenstrual age
  Prechtl's General Movement Assessment (GMA) is a clinical assessment tool that classifies writhing movements in preterm infants. Specifically, classification of writhing movements will be made as cramped synchronous, poor repertoire with cramped synchronicity, or poor repertoire.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Jantzie, PhD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kitase Y, Sato Y, Takahashi H, Shimizu M, Ishikawa C, Yamamoto H, Hayakawa M. A new type of swaddling clothing improved development of preterm infants in neonatal intensive care units. Early Hum Dev. 2017 Sep;112:25-28. doi: 10.1016/j.earlhumdev.2017.06.005. Epub 2017 Jul 1. PMID 28675824